CLINICAL TRIAL: NCT06595381
Title: Early Detection of Patients with Eating Disorders in General Practice
Status: Not yet recruiting | Type: Observational
Sponsor: Donini Lorenzo M (Other)
Responsible Party: Sponsor-Investigator, Donini Lorenzo M, MD, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: 0894/2023
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Eating Disorder Prevention; Eating Disorders
Keywords: Eating Disorder; Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder; general practice; prevention; early diagnosis
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to assess the efficacy of the Eating Disorder Proxy Screening Tool for General Practitioner (ED-PSTGP) as a tool for the early detection of eating disorders (EDs) in General Practice (GP). The ED-PSTGP is a hetero-evaluative questionnaire that investigates the presence of suspected eating disorder symptoms among the family members of the person completing the questionnaire. The study will involve adult patients over 18 years old enrolled in a general practice and their family members aged 16 years or older.

The main questions it aims to answer are:

* Can the ED-PSTGP questionnaire effectively identify patients with potential eating disorders through responses from a family member?
* How effective is the ED-PSTGP questionnaire in general practice as an early detection tool for eating disorders?

Participants will:

* Be asked by their General Practitioner (GP) to complete the ED-PSTGP questionnaire.
* If a positive result is found, invite the potentially affected family member to complete additional screening questionnaires online.

The potentially affected family member will be offered a teleconsultation with specialists and encouraged to contact the nearest reference center for ED treatment to further investigate potential eating disorders.

DETAILED DESCRIPTION:
Eating Disorders (EDs) represent a serious public health issue that, in recent years, has taken on the characteristics of a true social epidemic. Timely diagnosis and treatment play a crucial role in the resolution of the disorder and in the prevention of chronic complications. Unfortunately, many individuals seek care with significant delay, resulting in severe prognostic consequences and a high risk of chronicity. General Practitioners (GPs), as primary care providers in direct contact with the public, often represent the first point of contact between patients and the National Health System. The families of those affected by these disorders can play a crucial role in the diagnostic-therapeutic process by identifying the symptoms early, which may appear very subtle in the initial stages.

STUDY DESIGN Forty GPs, distributed across the national territory and selected by the Italian Society of Preventive Medicine and Lifestyle (SIMPeSV), will collaborate in the study. Enrollment will be non-competitive, and each participating GP will be required to administer the ED-PSTGP questionnaire to 30 adult patients.

The GP will be responsible for evaluating the test. The presence of a positive answer to any of the 13 items in the questionnaire will be considered sufficient to raise a suspicion of ED. Patients who complete a test evaluated as positive will be asked to provide the following questionnaires to the potentially affected family member:

* Eating Disorder Screen for Primary Care (ESP)
* Sick, Control, One stone, Fat, Food (SCOFF)
* Disordered Eating Questionnaire (DEQ)
* Beck Depression Inventory II (BDI II) The questionnaires and informed consent will be offered on an online platform and in Italian language.

The family members indicated as potentially affected by EDs will be offered a teleconsultation (with the operators from the Nutrition Science Research Unit of the University of Rome La Sapienza; and the Clinical Psychology and Counseling Service of the University of Rome La Sapienza) to further investigate the suspicion of eating disorder.

The GP will encourage individuals with suspected ED to contact the nearest reference center for ED treatment for diagnostic confirmation and possible management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, for patients enrolled by a General Practitioner (GP) to complete the ED-PSTGP questionnaire.
* Ability to provide informed consent for participation in the study.
* Age ≥ 16 years, for family members of GP patients, identified as pontentially affected by an eating disorder.

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (aged ≥18 years) enrolled by General Practitioners (GPs) across Italy and their family members aged ≥16 years. Patients are selected from GP practices to complete the ED-PSTGP questionnaire, which aims to identify potential cases of eating disorders (EDs). Family members identified by these patients as potentially affected by an ED will also be included in the study. All participants must be able to provide informed consent for participation and for the anonymized use of their data.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Predictive capacity of the Eating Disorder Proxy Screening Tool for General Practitioners (ED-PSTGP) questionnaire in identifying patients with EDs | 3 years from the start of participant enrollment.

SECONDARY OUTCOMES:
Efficacy of the ED-PSTGP questionnaire in General Practice as a tool for the early detection of individuals affected by EDs. | 3 years from the start of participant enrollment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Quaderni del Ministero della Salute n. 29, settembre 2017. Linee di indirizzo nazionali per la riabilitazione nutrizionale nei disturbi dell'alimentazione. www.quadernidellasalute.it.
- [Background] Steinhausen HC. The outcome of anorexia nervosa in the 20th century. Am J Psychiatry. 2002 Aug;159(8):1284-93. doi: 10.1176/appi.ajp.159.8.1284. PMID 12153817
- [Background] Qian J, Wu Y, Liu F, Zhu Y, Jin H, Zhang H, Wan Y, Li C, Yu D. An update on the prevalence of eating disorders in the general population: a systematic review and meta-analysis. Eat Weight Disord. 2022 Mar;27(2):415-428. doi: 10.1007/s40519-021-01162-z. Epub 2021 Apr 8. PMID 33834377
- [Background] Morgan JF, Reid F, Lacey JH. The SCOFF questionnaire: assessment of a new screening tool for eating disorders. BMJ. 1999 Dec 4;319(7223):1467-8. doi: 10.1136/bmj.319.7223.1467. No abstract available. PMID 10582927
- [Background] McNulty PA. Prevalence and contributing factors of eating disorder behaviors in active duty Navy men. Mil Med. 1997 Nov;162(11):753-8. PMID 9358723
- [Background] Luck AJ, Morgan JF, Reid F, O'Brien A, Brunton J, Price C, Perry L, Lacey JH. The SCOFF questionnaire and clinical interview for eating disorders in general practice: comparative study. BMJ. 2002 Oct 5;325(7367):755-6. doi: 10.1136/bmj.325.7367.755. No abstract available. PMID 12364305
- [Background] Lombardo C, Russo PM, Lucidi F, Iani L, Violani C. Internal consistency, convergent validity and reliability of a brief questionnaire on disordered eating (DEQ). Eat Weight Disord. 2004 Jun;9(2):91-8. doi: 10.1007/BF03325051. PMID 15330075
- [Background] Lombardo C, Cuzzolaro M, Vetrone G, Mallia L, Violani C. Concurrent validity of the Disordered Eating Questionnaire (DEQ) with the Eating Disorder Examination (EDE) clinical interview in clinical and non clinical samples. Eat Weight Disord. 2011 Sep;16(3):e188-98. doi: 10.1007/BF03325131. PMID 22290035
- [Background] Pinhas L, Morris A, Crosby RD, Katzman DK. Incidence and age-specific presentation of restrictive eating disorders in children: a Canadian Paediatric Surveillance Program study. Arch Pediatr Adolesc Med. 2011 Oct;165(10):895-9. doi: 10.1001/archpediatrics.2011.145. PMID 21969390
- [Background] Lahteenmaki S, Saarni S, Suokas J, Saarni S, Perala J, Lonnqvist J, Suvisaari J. Prevalence and correlates of eating disorders among young adults in Finland. Nord J Psychiatry. 2014 Apr;68(3):196-203. doi: 10.3109/08039488.2013.797021. Epub 2013 Jun 10. PMID 23750986
- [Background] Freund KM, Graham SM, Lesky LG, Moskowitz MA. Detection of bulimia in a primary care setting. J Gen Intern Med. 1993 May;8(5):236-42. doi: 10.1007/BF02600088. PMID 8505681
- [Background] Broomfield C, Stedal K, Touyz S, Rhodes P. Labeling and defining severe and enduring anorexia nervosa: A systematic review and critical analysis. Int J Eat Disord. 2017 Jun;50(6):611-623. doi: 10.1002/eat.22715. Epub 2017 Apr 25. English, Spanish. PMID 28444828
- [Background] Anstine D, Grinenko D. Rapid screening for disordered eating in college-aged females in the primary care setting. J Adolesc Health. 2000 May;26(5):338-42. doi: 10.1016/s1054-139x(99)00120-2. PMID 10775826